CLINICAL TRIAL: NCT06893744
Title: Effects of Different Occlusal Splints on Joint Vibrations in Bruxers
Brief Title: Effects of Different Occlusal Splints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Bora Akat, Assistant Professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 42/4
Record Dates: First submitted 2025-03-17; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2012-12

CONDITIONS: Bruxism; Bruxism, Sleep; Occlusal Splints
Keywords: Bruxism; Occlusal Splints; Bruxism, Sleep; TMJ
MeSH Terms: conditions — Bruxism; Sleep Bruxism | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blinded because they did not know the method of interventional treatment (occlusal splints) given to them. In addition, the outcome assessor was blinded because he assessed the patients with the occlusal splints out of their mouths. Therefore, this research had double blind study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Soft Splint (Experimental): It is a type of occlusal splint using soft material. It was applied to bruxist patients in accordance with the study design (Group 2).
  Interventions: Device: occlusal splint
- Hard Splint (Experimental): It is a type of occlusal splint using hard material. It was applied to bruxist patients in accordance with the study design (Group 3).
  Interventions: Device: occlusal splint
- Semi-soft Splint (Experimental): It is a type of occlusal splint using semi-soft material. They cover the advantages of soft and hard occlusal splints. It was applied to bruxist patients in accordance with the study design (Group 4).
  Interventions: Device: occlusal splint

INTERVENTIONS:
Device: occlusal splint

SUMMARY:
This study was carried out on 49 patients with bruxism and 15 asymptomatic individuals (group 1, control), totally 64 subjects. The selection of patients with bruxism was based on International Classification of Sleep Disorders Sleep bruxism diagnostic criteria. 16 patients were treated with soft splint (group 2), 17 patients were treated with hard splint (group 3) and left 16 patients were treated with semi-soft splint (group 4). Joint vibration records were made with JVA (Biopak system BioResearch , Inc., Milwaukee, WI) device during the opening and closing movements. The recordings were made before and after occlusal splint treatment for three months in patients with bruxism. The recordings of individuals in control group was made two times at three months intervals. Also clinical evaluation was made with questionnaire forms. The study was approved by the ethical committee and each subject gave informed consent.

DETAILED DESCRIPTION:
It was demonstrated that occlusal splints are effectual on improving clinical symptoms and reducing patient complaints in patients with bruxism. However the effects of occlusal splints on joint vibrations are not fully elucidated. The aim of this study is to evaluate the effects of three different occlusal splints (soft, hard and semi-soft) on joint vibrations in patients with bruxism and to compare with asymptomatic individuals. And also clinical symptoms and patient complaints were evaluated with questionnaire forms.

This study was carried out on 49 patients with bruxism and 15 asymptomatic individuals (group 1, control), totally 64 subjects. The selection of patients with bruxism was based on International Classification of Sleep Disorders Sleep bruxism diagnostic criteria. 16 patients were treated with soft splint (group 2), 17 patients were treated with hard splint (group 3) and left 16 patients were treated with semi-soft splint (group 4). Joint vibration records were made with JVA (Biopak system BioResearch , Inc., Milwaukee, WI) device during the opening and closing movements. The recordings were made before and after occlusal splint treatment for three months in patients with bruxism. The recordings of individuals in control group was made two times at three months intervals. Also clinical evaluation was made with questionnaire forms. The study was approved by the ethical committee and each subject gave informed consent.

There was no significant difference in joint vibration parameters between patients with bruxism and asymptomatic individuals before treatment (p>0.0063). Between the increase in soft group and reduction respectively in hard group and semi-soft group for total integral values variations, after treatment at the opening movement for left joint were statistically significant (p=0.005 and p<0.001). Total integral, i>300 Hz, i<300 Hz, Peak amplitude, Peak frequency values of patients with bruxism were observed to be higher than the value of asymptomatic individuals, allthough there was no statistical difference. After three different occlusal splint treatment, it was observed that there was clinically improvement in patient complaints.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a complaint of grinding/clenching during sleep
* One or more of the following occurs:

  1. abnormal wear of the teeth
  2. sounds associated with the bruxism
  3. jaw muscle discomfort
* No other medical or mental disorders that affecting masticatory muscles activity

Exclusion Criteria:

* Patients with missing at least 2 posterior teeth, except for the third molars
* Presence of Myofascial Pain Dysfunction (MPD)
* Presence of major neurological, psychiatric or motor disorders
* Patients using medications, influencing sleep or motor functions
* Patients with alcohol or drug addiction
* Patients ongoing any dental treatment
* Patients using occlusal splint or exposing the treatment for TMJ disorders in the last 3 months.
* Patients with pregnancy
* Patients with cancer
* Patients with scheduled surgery operation
* Patients with pericoronitis or supraeruption of 3rd molar

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2013-02-15 (Actual); Study Completion 2014-08-15 (Actual)

PRIMARY OUTCOMES:
Vibration analysis resulting from the movement between temporomandibular joint surfaces with JVA (Joint Vibration Analysis) device | 3 days
  Joint vibration analysis resulting from the movement between temporomandibular joint surfaces was performed by using a Joint Vibration Analysis device (BioPAK (BioResearch, Inc., Milwaukee, WI). Joint vibration analysis parameters were evaluated after occlusal splint treatments in patients with bruxism for each arm.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Akat B, Akoren AC, Tamam E. Effects of Different Occlusal Splints on Joint Vibrations in Bruxers. Medicina (Kaunas). 2025 Jun 12;61(6):1083. doi: 10.3390/medicina61061083. PMID 40572771